CLINICAL TRIAL: NCT06547346
Title: To Evaluate the Acceptability and Palatability of a Hypoallergenic Nutritionally Complete Powdered Amino Acid Formula With HMO (Human Milk Oligosaccharides) for the Dietary Management of Cows' Milk Allergy (CMA) and Multiple Food Protein Allergies (MFPA) in Children Over ≥1 Year.
Brief Title: Acceptability and Palatability Study of Paediatric Amino Acid Feed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AJ2022
Record Dates: First submitted 2024-04-25; First posted 2024-08-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients well established on tube feeds will act as their own control (Experimental)
  Interventions: Dietary Supplement: Alfamino Junior

INTERVENTIONS:
Dietary Supplement: Alfamino Junior — To recruit 15 children and evaluate the acceptability (including gastrointestinal tolerance), palatability and compliance of a hypoallergenic amino acid powdered formula (neutral and vanilla flavours) with HMO's for the dietary management of presumed cows' milk allergy, multiple food protein allergies and other conditions where an amino acid formula is recommended in children ≥1 year of age.

SUMMARY:
Product acceptability and palatability data from a minimum of 15 participants are required to submit an application to the Advisory Committee on Borderline Substances (ACBS) and the Health Service Executive (HSE) for Ireland for product registration

DETAILED DESCRIPTION:
The study product, Alfamino Junior (neutral or vanilla flavour) is a is a food for special medical purposes, as defined by EU Regulation No 609/2013, ACBS approved, prescribable on FP10 (GP10 in Scotland).

Alfamino Junior (neutral or vanilla flavour) is is for complete nutritional support of children ≥1 year with cows' milk allergy, multiple food allergies and other conditions where an amino acid formula is recommended.

This is an open label nonrandomised acceptability, palatability and compliance study to evaluate the tolerance of the study formulas in 15 children.

Palatability is recorded over a 7day study period, acceptability is recorded days 1-7 and days 22-28 of the study period, with patient compliance recorded over the full 28 day study period

ELIGIBILITY:
Inclusion criteria:

* Children ≥1 year of age who require an amino acid-based formula (ideally already established on Alfamino or another amino acid formula dependent on feasibility of reaching required numbers or currently on a plant-based milk and need extra nutrition from an amino acid formula) for the dietary management of presumed CMA, or multiple food allergies and other conditions where an amino acid formula is recommended
* All children ≥1 year of age where they are consuming either orally or via a tube 200mls or more of amino acid formula.
* Children with the ability to indicate palatability of the formula (NB there will be simple symbols to help young children and nonverbal children indicate whether the formula is palatable). If an infant is tube fed if they are able to have tastes orally.
* Willingly given, written, informed consent from patient or parent/guardian.

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator.
* Children less than 1 year of age
* Children with significant renal or hepatic impairment
* Change in current medication or use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator e.g. thickener, PPIs etc (must be recorded in patient case record file).
* Participation in another intervention study within 2 weeks of this study.
* Caregiver unable to read and write in English (will need to complete 1 month of forms at home on behalf of participants).

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Number of children reporting gastrointestinal tolerance using an online questionnaire. | 7 days
  Number of patients reporting diarrhoea and / or constipation, Bloating and / or distension, Nausea and / or vomiting, Burping / flatulence / regurgitation, Abdominal discomfort/ pain, measured as symptoms and graded as none, mild moderate or severe
Palatability, indicated via symbols of how much the product is liked using online questionnaire. | 7 days
  Number of children who like the appearance, taste, smell graded as as 5 likert scale of an online questionnaire from really liked to really did not like using happy to sad images to correctly identify outcome.
Participant compliance | 7 days
  How many feeds and volume prescribed each day, How many feeds and volume taken

CONTACTS AND LOCATIONS:
Locations (1):
- Paediatric allergy, Leeds Children's Hospital, Clarendon Wing, Leeds General Infirmary, Leeds,, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided